CLINICAL TRIAL: NCT01930786
Title: ASPIRE: Adult SPasticity International REgistry on BOTOX® Treatment
Brief Title: An Adult Spasticity Registry of OnabotulinumtoxinA Treatment
Acronym: ASPIRE
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-BTX-SP-12-001
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- onabotulinumtoxinA: onabotulinumtoxinA administered according to physician standard of care. All treatment decisions lie with the physician.
  Interventions: Drug: onabotulinumtoxinA

INTERVENTIONS:
Drug: onabotulinumtoxinA — onabotulinumtoxinA administered according to physician standard of care. All treatment decisions lie with the physician.
  Other Names: BOTOX®; botulinum toxin Type A

SUMMARY:
This is a registry study in adults with spasticity to determine onabotulinumtoxinA use in clinical practice. Treatment will be administered in accordance with physician standard practice. All treatment decisions lie with the physician.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with onabotulinumtoxinA according to the decision of the physician for spasticity
* Willingness to complete study questionnaires and answer study questions by phone or internet

Exclusion Criteria:

* Concurrent participation in a clinical trial for spasticity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Muscle Spasticity
Sampling Method: Non-Probability Sample
Enrollment: 744 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients Reporting Satisfaction with Treatment | 5 Weeks
Percentage of Health Care Providers Reporting Satisfaction with Treatment | 12 Weeks

SECONDARY OUTCOMES:
Physical Functioning on a 5-Point Scale | 5 Weeks
Severity of Pain on an 11-Point Scale | 5 Weeks
Disability Assessment on a 4-Point Scale | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aleks Zuzek, Study Director — Allergan
Locations (55):
- United States (26):
  - Loma Linda University School Of Medicine, Loma Linda, California
  - MS Center of California, Newport Beach, California
  - Sutter Health General Hospital, Sacramento, California
  - Design Neuroscience Center, Doral, Florida
  - Brooks Rehabilitation Hospital, Jacksonville, Florida
  - Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - Gil, Ramon A., Port Charlotte, Florida
  - Kernan Hospital, Baltimore, Maryland
  - MedTechnical, PLLC, Silver Spring, Maryland
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - The Curators of the University of Missouri on behalf of University of Missouri Health Care, Columbia, Missouri
  - Seacoast Physiatry, Exeter, New Hampshire
  - CentraState Medical Center, Freehold, New Jersey
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Dayton Center for Neurological Disorders, Dayton, Ohio
  - Albert Einstein Healthcare Network, Moss Rehabilitation Hospital, Elkins Park, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn Medicine Rittenhouse, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Metrolina Neurological Assoc., PA, Rock Hill, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Memorial Hermann Hospital, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Swedish Neuroscience Institute, Seattle, Washington
  - Center for Neurological Disorders, S.C., Milwaukee, Wisconsin
- France (5):
  - Hôpital Morvan, Brest, Finistere
  - Pôle Saint Helier, Rennes, Ille Et Vilaine
  - CHU de Grenoble - Hôpital Sud, Échirolles, Isere
  - Hopital Saint Philibert - GHICL Lille, Lomme, Nord
  - Centre Hospitalier de Pau, Pau, Pyrenees Atlantiques
- Germany (6):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
  - Universitaetsklinikum Jena, Jena, Thuringia
  - Parkinson Klinik Wolfach GmbH & Co KG, Baden Wuerttemberg
- Italy (4):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero - Universitaria Maggiore delle Carità, Novara
  - Policlinico Universitario Agostino Gemelli, Roma
- Spain (7):
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital de Conxo (Santiago de Compostela) GALICIA, Santiago de Compestela, Pontevedra
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Institut de Recerca-VHIR, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Complejo Hospitalario de Pontevedra, Pontevedra
- Taiwan (2):
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- United Kingdom (5):
  - The National Hospital for Neurology & Neurosurgery, London, Greater London
  - Birch Hill Hospital, Rochdale, Greater Manchester
  - Kent and Canterbury Hospital, Kent, Kent
  - The Walton Centre, Liverpool, Merseyside
  - Nottingham University Hospitals City Campus, Nottingham, Nottinghamshire

REFERENCES:
- [Derived] Wissel J, List C, Schwartz M, Nelson M, Musacchio T, Duarte E. Relief of pain associated with spasticity in adult patients after treatment with onabotulinumtoxinA: Post hoc observational results from the ASPIRE study. PM R. 2025 Sep 30. doi: 10.1002/pmrj.70013. Online ahead of print. PMID 41025675
- [Derived] Bavikatte G, Francisco GE, Jost WH, Baricich A, Duarte E, Tang SFT, Schwartz M, Nelson M, Musacchio T, Esquenazi A. Pain, disability, and quality of life in participants after concurrent onabotulinumtoxinA treatment of upper and lower limb spasticity: Observational results from the ASPIRE study. PM R. 2024 Nov;16(11):1175-1189. doi: 10.1002/pmrj.13195. Epub 2024 May 30. PMID 38813838
- [Derived] Bavikatte G, Esquenazi A, Dimyan MA, Dashtipour K, Feng W, Mayadev A, Fanning K, Musacchio T, Zuzek A, Francisco GE. Safety and Real-World Dosing of OnabotulinumtoxinA for the Treatment of Adult Spasticity: Post Hoc Analysis of the Adult Spasticity International Registry Study. Am J Phys Med Rehabil. 2024 Jul 1;103(7):580-587. doi: 10.1097/PHM.0000000000002410. Epub 2024 Jan 8. PMID 38206635
- [Derived] Esquenazi A, Francisco GE, Feng W, Baricich A, Gallien P, Fanning K, Zuzek A, Bandari DS, Wittenberg GF. Real-World Adherence to OnabotulinumtoxinA Treatment for Spasticity: Insights From the ASPIRE Study. Arch Phys Med Rehabil. 2021 Nov;102(11):2172-2184.e6. doi: 10.1016/j.apmr.2021.06.008. Epub 2021 Jul 7. PMID 34245684
- [Derived] Esquenazi A, Bavikatte G, Bandari DS, Jost WH, Munin MC, Tang SFT, Largent J, Adams AM, Zuzek A, Francisco GE. Long-Term Observational Results from the ASPIRE Study: OnabotulinumtoxinA Treatment for Adult Lower Limb Spasticity. PM R. 2021 Oct;13(10):1079-1093. doi: 10.1002/pmrj.12517. Epub 2021 Jan 11. PMID 33151636
- [Derived] Francisco GE, Jost WH, Bavikatte G, Bandari DS, Tang SFT, Munin MC, Largent J, Adams AM, Zuzek A, Esquenazi A. Individualized OnabotulinumtoxinA Treatment for Upper Limb Spasticity Resulted in High Clinician- and Patient-Reported Satisfaction: Long-Term Observational Results from the ASPIRE Study. PM R. 2020 Nov;12(11):1120-1133. doi: 10.1002/pmrj.12328. Epub 2020 Feb 27. PMID 31953896